CLINICAL TRIAL: NCT05136586
Title: Effects of Two Stress Management Procedures on Performances During Objective Structured Clinical Examination (OSCE) for Medical Students : Relaxing Breathing Combined With Biofeedback or Meditative Stimulation : ECOSTRESS Study
Brief Title: Effects of Relaxing Breathing With Biofeedback or Meditative Stimulation on Performances During OSCE of Medical Students
Acronym: ECOSTRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, Principal Investigator, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ECOSTRESS
Record Dates: First submitted 2021-11-04; First posted 2021-11-29 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Stress, Psychological; Stress, Physiological; Exam Stress; Performance Anxiety; Rumination
Keywords: Stress management and performance; Medical education
MeSH Terms: conditions — Stress, Psychological; Rumination Syndrome | interventions — Biofeedback, Psychology; Meditation

STUDY DESIGN:
Intervention Model Description: 4 parallels groups
Who Masked: Investigator, Outcomes Assessor
Masking Description: Performance is evaluated by assessors who are blind to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Biofeedback (Experimental): Relaxing breathing exercise coupled with biofeedback before the circuit, no intervention after
  Interventions: Other: Biofeedback
- Meditation (Experimental): Meditative stimulation audio tape before the circuit, no intervention after
  Interventions: Other: Meditation
- Control and biofeedback post OSCE (Experimental): Standardised video before the circuit, Relaxing breathing exercise coupled with biofeedback after the OSCE
  Interventions: Other: Control and biofeedback post OSCE
- Control and control post OSCE (Sham Comparator): Standardised video before the circuit, no intervention after
  Interventions: Other: Control and control post OSCE

INTERVENTIONS:
Other: Biofeedback — 6 minutes of relaxing breathing exercise coupled with hert rate variability biofeedback guided on eMWave Pro software on a computer just before entering the examination circuit.
  After the circuit, 6 minutes of free activity where the participants will not be given any instruction.
  Other Names: Relaxing breathing exercise coupled with biofeedback before the circuit, no intervention after
  Arms: Biofeedback
Other: Meditation — 6 minutes of listening an audio tape made for the study that inspire mindfulness like meditation associated with psychological stimulation (positive encouragement) just before entering the examination circuit.
  After the circuit, 6 minutes of free activity where the participants will not be given any instructions.
  Other Names: Meditative stimulation audio tape before the circuit, no intervention after
  Arms: Meditation
Other: Control and biofeedback post OSCE — 6 minutes of standardised neutral video on general topics that generates no modification of affects just before entering the examination circuit.
  After the circuit, 6 minutes of relaxing breathing exercise coupled with hert rate variability biofeedback guided on eMWave Pro software on a computer
  Other Names: Standardised video before the circuit, relaxing breathing exercise coupled with biofeedback after
  Arms: Control and biofeedback post OSCE
Other: Control and control post OSCE — 6 minutes of standardised neutral video on general topics that generates no modification of affects just before entering the examination circuit.
  After the circuit, 6 minutes of of free activity where the participants will not be given any instruction.
  Other Names: Standardised video before the circuit, no intervention after
  Arms: Control and control post OSCE

SUMMARY:
Objective Structured Clinical Examination (OSCE) is a newly implemented evaluation standard for medical student and is a determinant part of the national competition they have to undergo.

Medical studies, especially during examen period, are significantly associated with risk of developping depressions or anxious trouble, wich led to lesser performance, impaired memorization and impaired workload capacities.

Relaxation breathing techniques coupled with heart rate variability (HRV) biofeedback and meditation are procedures used to reduce the stress level.

There is currently no study on the effect of stress management procedures on the performance during OSCE for medical student.

DETAILED DESCRIPTION:
This randomized, controlled, monocentric study will take place during mandatory rehearsal of Objective Structured Clinical Examination for third year medical student. For examination purpose, the students will be divided in four groups that will undergo identical exam in the same time in four parallels circuits.

Before entering the circuit, all the students will received information for the study and sign consent.

All the students will be equipped with emWAve® devices that allows us to collect heart rate variability as physiological stress marker during the time of the intervention. Participants will undergo short questionnaires regarding perceived stress.

Then the groups of students will be randomized in four interventions groups for receiving a combination of intervention before and/or after the examination circuit. All the interventions last six minutes long. The randomisation groups are :

* Relaxing breathing exercise coupled with biofeedback before the circuit, no intervention after
* Meditative stimulation audio tape before the circuit, no intervention after
* Standardised video as controlled group before the circuit and a relaxing breathing exercise coupled with biofeedback after
* Standardised video as controlled group before and not intervention after

At the end of the examination circuit, all the students will undergo short questionnaires regarding stress, participants will get equipped with emWAve ® devices again and participants will get the second intervention depending on the randomisation group.

Main objective is to show that relaxing breathing exercise coupled with biofeedback or meditative stimulation is better than an standardised video on performance during OSCE.

The main outcome is student grade at the exam, as determined by university evaluator who is blind to the intervention and with no links to the study.

Secondary objectives are to compare the effects of the interventions on measured physiological stress, psychological stress, and negative rumination.

ELIGIBILITY:
Inclusion Criteria:

* Adult person
* Registered as medical student at the university
* Participating at OSCE examination
* Have signed an informed consent form.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Differences in Performance | During the first 2 hours of the inclusion
  The performance is student grade at the exam, as determined by university evaluator

SECONDARY OUTCOMES:
Differences of Physiological stress | During the first 2 hours of the inclusion
  Heart rate variation collected by emWave® devices
Differences of Psychological stress | Four times : before first intervention, before OSCE circuit, just after OSCE circuit, just after second intervention
  Numerical Visual analog scales (VAS) on perceived stress from zero to 100: maximum Numerical VAS on resourcefulness nedeed an avalaible perceived from zero to maximum
Difference of Resourcefulness | Four times : before first intervention, before OSCE circuit, just after OSCE circuit, just after second intervention
  Numerical VAS on resourcefulness needeed an available perceived from zero to 100: maximum
Characterisation of stress | Four times : before first intervention, before OSCE circuit, just after OSCE circuit, just after second intervention
  Numerical VAS on characterisation of stress perceived from negative to positive
Differences of Self confidence | Four times : before first intervention, before OSCE circuit, just after OSCE circuit, just after second intervention
  Numerical VAS on self confidence perceived from zero to 100: maximum
Differences of Psychological stress consequences | Three times : before first intervention, before OSCE circuit, just after second intervention
  Activation-Deactivation Adjective Check List: for the four subscales: Energy, Tiredness, Tension , and Calmness
Differences of Ruminations | Just after second intervention at the end of the OSCE
  Brief rumination scale questionnaire
Individual psychological characteristics | Just after second intervention at the end of the OSCE
  Personality traits (Big-5)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Rode, M.D., Ph.D., Study Chair — Claude Bernard University
Locations (1):
- Marc lilot, Lyon, France

REFERENCES:
- [Derived] Le Saux O, Canada B, Debarnot U, Haouhache NEH, Lehot JJ, Binay M, Cortet M, Rimmele T, Duclos A, Rode G, Lilot M, Schlatter S. Association of Personality Traits With the Efficacy of Stress Management Interventions for Medical Students Taking Objective Structured Clinical Examinations. Acad Med. 2024 Jul 1;99(7):784-793. doi: 10.1097/ACM.0000000000005714. Epub 2024 Mar 25. PMID 38534105